CLINICAL TRIAL: NCT00083967
Title: A Randomized, Double-Masked, Placebo Controlled, Parallel Group, Multi-Center, Dose-Ranging Study of Denufosol Tetrasodium (INS37217) Intravitreal Injection in Subjects With Rhegmatogenous Retinal Detachment
Brief Title: Study of Denufosol (INS37217) in Subjects With Rhegmatogenous Retinal Detachment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-102
Record Dates: First submitted 2004-06-03; First posted 2004-06-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Retinal Detachment
Keywords: rhegmatogenous retinal detachment; detached retina; retinal tear; retinal break
MeSH Terms: conditions — Retinal Detachment; Retinal Perforations | interventions — denufosol tetrasodium; Intravitreal Injections

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Intravitreal Injection

SUMMARY:
The purpose of this study is to test if denufosol will remove the fluid build-up in the eye so that the retina can be re-attached without invasive surgery.

DETAILED DESCRIPTION:
The purpose of this trial is to determine if administration of denufosol is well-tolerated and more efficacious than placebo in stimulating subretinal fluid reabsorption and retinal reattachment without surgical intervention in subjects presenting with rhegmatogenous retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* have rhegmatogenous retinal detachment in only one eye
* be able to receive intravitreal injection of study drug and be able to wait 24(+/- 6) hours to have detachment surgically treated or retinal breaks repaired per judgement of investigator
* no more than 3 separate identifiable retinal breaks that are clustered together and confined within an area no more than 2 clock hours in extent
* retinal detachment must be large enough such that it cannot be immediately repaired with laser photocoagulation or cryotherapy
* have pinhole acuity (using ETDRS) of macula-on, 20/50 or better in both eyes OR macula-off, 20/50 or better in non-study eye and have history, prior to detachment, of reading capability in study eye

Exclusion Criteria:

* have a non-rhegmatogenous retinal detachment
* have large retinal break(s) whose total break area is greater than 1 clock hour in extent
* have evidence of atrophic retinal pigment epithelium, choroid, choroidal detachment or intraocular inflammation
* be monocular
* have a prior retinal detachment repair or a congenital condition that places a greater risk for rhegmatogenous retinal detachment
* have proliferative vitreoretinopathy greater than grade B
* have pre-existing subretinal or vitreous hemorrhage, corneal opacity, or other conditions which limit the view of peripheral retina
* have any co-existing macular pathology or other retinal conditions that can limit visual acuity
* currently have uncontrollable elevated intraocular pressure, advanced glaucoma, or any history or current evidence of endophthalmitis in the affected eye
* have symptoms consistent with a rhegmatogenous retinal detachment such as visual disturbance greater than 14 days prior to screening if macula-on OR history of loss of reading vision in affected eye for greater than 6 days prior to screening if macula-off
* have a retinal detachment with evidence of demarcation lines or evidence of subretinal fibrosis visible upon fundus examination
* be currently taking medications that could obscure or confound study results including acetazolamide (Diamox) and dorzolamide
* have had a periocular, retrobulbar or intravitreal injection in the affected eye, including corticosteroids in the 3 months prior to screening or require one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Compare safety and tolerability of single and/or multiple intravitreal injections of three dose levels of denufosol vs. placebo
Compare efficacy of denufosol vs. placebo as a treatment for detachment of the retina in RRD subjects

SECONDARY OUTCOMES:
Identify one or more dose levels of denufosol as safe and potentially effective to warrant study in Phase 3
Evaluate utility of 3D B-scan ultrasound technology as endpoint for objectively describing volume of retinal detachment

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director
Locations (33):
- United States (33):
  - Retina Center, P.C., Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Vitreous Associates Medical Group, Los Angeles, California
  - Retina Consultants San Diego, Poway, California
  - Danbury Eye Physicians & Surgeons, P.C., Danbury, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Central Florida Retina, Orlando, Florida
  - The University of Chicago, Chicago, Illinois
  - Illinois Retina Associates, S.C., Joliet, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - University of Kentucky, The Kentucky Clinic, Lexington, Kentucky
  - Maine Vitreoretinal Consultants, Bangor, Maine
  - National Retina Institute, Chevy Chase, Maryland
  - New England Eye Center, Boston, Massachusetts
  - Kresge Eye Institute/Hutzel Hospital, Detroit, Michigan
  - Retina Associates, Kansas City, Missouri
  - Retina Associates of NJ, Millburn, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - Retina Associates of NJ, Wayne, New Jersey
  - NY Eye and Ear Infirmary, New York, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Retina Assocites of Cleveland, Inc., Cleveland, Ohio
  - Cleveland Clinical Foundation, Cleveland, Ohio
  - Retina Associates of Cleveland, Lakewood, Ohio
  - Retina Associates of Cleveland, Lorain, Ohio
  - Retina Associates of Cleveland, Middleburg Heights, Ohio
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Austin Retina, Austin, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Wagner Mandell Retina Center, Norfolk, Virginia
  - Wagner Mandell Retina Center, Virginia Beach, Virginia
  - Medical College of Wisconsin/The Eye Institute, Milwaukee, Wisconsin